CLINICAL TRIAL: NCT04757675
Title: A Comparison of S-ketamin, Dexmedetomidine, and Combination as Premedication in Children Undergoing ENT Surgery
Brief Title: S-ketamin Premedication in Pediatric EENT Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Hui Qiao, Clinical Anesthesiologist, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Premedication s-ketamin
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Emotions; Separation Anxiety; Pain, Procedural
MeSH Terms: conditions — Anxiety, Separation; Pain, Procedural | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.3 SK iv (Experimental): 0.3 μg/kg intravenous injection s-ketamin
  Interventions: Drug: S-ketamine 0.3
- 0.5 SK iv (Experimental): 0.5 μg/kg intravenous injection s-ketamin
  Interventions: Drug: S-ketamine 0.5
- 2 SK in (Experimental): 2 μg/kg intranasal s-ketamin
  Interventions: Drug: S-ketamine 2
- 1 SK in + 1 DEX in (Experimental): 1 μg/kg intranasal s-ketamin + 1 μg/kg intranasal dexmedetomidine
  Interventions: Drug: S-ketamine 1+Dexmedetomidine 1
- 0.5 SK in + 2 DEX in (Experimental): 0.5 μg/kg intranasal s-ketamin + 2 μg/kg intranasal dexmedetomidine
  Interventions: Drug: S-ketamine 0.5 +Dexmedetomidine 2

INTERVENTIONS:
Drug: S-ketamine 0.3 — 0.3 μg/kg intravenous injection s-ketamin
  Other Names: Jiangsu Hengrui Medicine Co.,Ltd.
  Arms: 0.3 SK iv
Drug: S-ketamine 0.5 — 0.5 μg/kg intravenous injection s-ketamin
  Other Names: Jiangsu Hengrui Medicine Co.,Ltd.
  Arms: 0.5 SK iv
Drug: S-ketamine 2 — 2 μg/kg intranasal s-ketamin
  Other Names: Jiangsu Hengrui Medicine Co.,Ltd.
  Arms: 2 SK in
Drug: S-ketamine 1+Dexmedetomidine 1 — 1 μg/kg intranasal s-ketamin + 1 μg/kg intranasal dexmedetomidine
  Other Names: Jiangsu Hengrui Medicine Co.,Ltd.
  Arms: 1 SK in + 1 DEX in
Drug: S-ketamine 0.5 +Dexmedetomidine 2 — 0.5 μg/kg intranasal s-ketamin + 2 μg/kg intranasal dexmedetomidine
  Other Names: Jiangsu Hengrui Medicine Co.,Ltd.
  Arms: 0.5 SK in + 2 DEX in

SUMMARY:
We aim to investigate the effects of premedication (intranasal or intravenous administration) of s-ketamin, dexmedetomidine, and combination for premedication in children undergoing ENT surgery.

DETAILED DESCRIPTION:
Three hundred children aged between 2 and 12 years were randomly allocated to one of five groups: 0.3 μg/kg intravenous injection s-ketamin; 0.5 μg/kg intravenous injection s-ketamin; 2 μg/kg intranasal s-ketamin group; 1 μg/kg intranasal s-ketamin + 1 μg/kg intranasal dexmedetomidine group; 0.5 μg/kg intranasal s-ketamin + 2 μg/kg intranasal dexmedetomidine group.

The modified Yale Preoperative Anxiety Scale (m-YPAS) was used to assess preoperative anxiety at 1, 5, 10, 20, and 30min after premedication. A 4-point emotional state score was used to evaluate participators when they were separated from their parents and their response to intravenous cannulation or facemask application. Agitation scores (Pediatric Anesthesia Emergence Delirium [PAED] scale) and POV was assessed in the postanesthetic care unit (PACU). Times to endotracheal tube or laryngeal mask airway removal, discharge from the PACU, and patients' satisfaction degree were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* After obtaining the informed consent from their parents or proxies, the children aged 2 to 12 years, scheduled for elective ENT surgery, of American Society of Anesthesiologists (ASA) I or II were enrolled in this study.

Exclusion Criteria:

* Congenital heart diseases, congenital dysplasia, obstructive sleep apnea syndrome, upper respiratory tract infection, body mass index (BMI) ≥25, allergy to S-ketamin or dexmedetomidine, and severe liver or kidney disease.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The modified Yale Preoperative Anxiety Scale | 1 min after premedication
  A validated observational tool for assessing children's anxiety
The modified Yale Preoperative Anxiety Scale | 5 min after premedication
  A validated observational tool for assessing children's anxiety
The modified Yale Preoperative Anxiety Scale | 10 min after premedication
  A validated observational tool for assessing children's anxiety
The modified Yale Preoperative Anxiety Scale | 20 min after premedication
  A validated observational tool for assessing children's anxiety
The modified Yale Preoperative Anxiety Scale | 30 min after premedication
  A validated observational tool for assessing children's anxiety

SECONDARY OUTCOMES:
Parental Separation Anxiety Scale (PSAS) | 30 min after premedication
  1. = easy separation
  2. = whimpers, but is easily reassured, not clinging
  3. = cries and cannot be easily reassured, but not clinging to parents
  4. = crying and clinging to parents
Emotional State Scale | 15 min after premedication
  Successful venous cannulation was defined as an ESS-4 ≤2 at the time of attempted cannulation, regardless of whether the vein was actually cannulated on the first attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qiao, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Derived] Qiao H, Zhuang Y, Lv P, Ye Z, Lu Y, Jia J. Intranasal esketamine versus esketamine-dexmedetomidine combination for premedication in pediatric patients undergoing strabismus surgery: a randomized controlled trial. Transl Pediatr. 2024 Aug 31;13(8):1327-1335. doi: 10.21037/tp-24-45. Epub 2024 Aug 28. PMID 39263280